CLINICAL TRIAL: NCT03814330
Title: A Comparison of Two Different Anesthetic Application (Sedation / Analgesia & LMA) on Anxiety Level and Patient Satisfaction in Patients With in Vitro Fertilization: Prospective Randomized Clinical Trial
Brief Title: A Comparison of Sedation/Analgesia & LMA on Anxiety Level and Patient Satisfaction in In-Vitro Fertilization
Acronym: IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof. Dr. Sedat Akbas, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: sedatakbas5
Record Dates: First submitted 2019-01-04; First posted 2019-01-24 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia; In-vitro Fertilization; Analgesia
Keywords: Anesthesia management; In-vitro Fertilization; Sedation-Analgesia
MeSH Terms: conditions — Agnosia | interventions — Analgesia; Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation/Analgesia (Placebo Comparator): Patients with applied sedation analgesia will perform State-Trait Anxiety Inventory and Quality of Recovery Score
  Interventions: Diagnostic Test: State-Trait Anxiety Inventory; Diagnostic Test: Quality of Recovery Score; Other: Sedation/Analgesia
- Laryngeal Mask Airway (Active Comparator): Patients with applied Laryngeal Mask Airway will perform State-Trait Anxiety Inventory and Quality of Recovery Score
  Interventions: Diagnostic Test: State-Trait Anxiety Inventory; Diagnostic Test: Quality of Recovery Score; Device: Laryngeal Mask Airway

INTERVENTIONS:
Diagnostic Test: State-Trait Anxiety Inventory — State-Trait Anxiety Inventory measures state anxiety levels and is an easy-to-implement inventory that the individual can answer on his/her own. State-Trait Anxiety Inventory determines how the individual feels himself / herself at a given moment and under certain conditions. It is widely used in preoperative anxiety measurement
Diagnostic Test: Quality of Recovery Score — Recovery Quality Score-40 (Quality of Recovery Score) and is used to measure the quality of postoperative recovery. This form consists 40 items and is divided into 5 subgroups according to various aspects of the improvement. There are a total of 40 items, 9 related to emotional state, 12 related to physical comfort, 7 related to psychological support, 5 related to physical independence and 7 items related to pain. The questionnaire is scored as a minimum of 40 to a maximum of 200.
  Other Names: Recovery Quality Score-40
Other: Sedation/Analgesia — Patients will be performed the procedure with sedation/analgesia under the condition of spontaneous breathing.
  Arms: Sedation/Analgesia
Device: Laryngeal Mask Airway — Patients will be performed the procedure with Laryngeal Mask Airway during the procedure. Laryngeal Mask Airway is a supraglottic airway device to ventilate the patients during anesthetic procedure.
  Arms: Laryngeal Mask Airway

SUMMARY:
In vitro fertilization (IVF) is a new expertise of our age. Anesthesia during the assisted reproduction technique is usually required during oocyte removal, which is one of the basic steps throughout the entire procedure. Until now, different anesthetic techniques such as conscious sedation, general anesthesia and regional anesthesia have been tried, no superiority has been proved against each other. The main point of anesthesia management in IVF is to minimize anesthesia exposure to avoid harmful effects on embryo division and fertilization.

The aim of this prospective randomized clinical trial was to compare two different anesthesia applications (sedation & laryngeal mask airway) on anxiety and patient satisfaction in patients with IVF.

DETAILED DESCRIPTION:
In vitro fertilization (IVF) is a new expertise of our age. Anesthesia during the assisted reproduction technique is usually required during oocyte removal, which is one of the basic steps throughout the entire procedure. Until now, different anesthetic techniques such as conscious sedation, general anesthesia and regional anesthesia have been tried, no superiority has been proved against each other. The main point of anesthesia management in IVF is to minimize anesthesia exposure to avoid harmful effects on embryo division and fertilization.

IVF requires the collection of mature oocytes from the ovaries of infertile patients. These oocytes are then fertilized in vitro and allowed to become embryos. Afterwards, these embryos are transferred into the uterus of the patients. Ultrasonography-guided transvaginal aspiration makes oocyte intake less invasive compared to prior techniques and can be administered within 30 minutes. With the development of this method, trauma was minimalized and side effects were reduced. However, the possible effects of different anesthetics on oocytes are still being discussed. The potential side effects of different anesthesia applications have been observed not only in patients receiving oocytes, but also in embryo development and pregnancy success due to the quality of oocytes. The pain of patients is common after the puncture of the vaginal fornix. It is usually defined as deep menstrual pain, quickly disappears and leaves a mild abdominal pain. Therefore, the anesthetist should perform adequate pain relief to immobilize the patient to avoid the risk of perforating the vessels during the procedure. Another challenge for the anesthesiologist is to alleviate the increased anxiety associated with social and psychological stress associated with IVF.

Anxiety may develop before and after the procedure, especially in patients undergoing oocyte collection. The patient's anxiety is usually present before entering the operating room. The assessment, which was started to be developped by investigators, was aimed to measure state anxiety levels in normal and non-normal individuals. State-Trait Anxiety Inventory measures state anxiety levels and is an easy-to-implement inventory that the individual can answer on his/her own. The State Anxiety Scale determines how the individual feels himself / herself at a given moment and under certain conditions. It is widely used in preoperative anxiety measurement.

Patient satisfaction depends on the patient's expectations and the benefits expected by the patients with the service they receive. Patient satisfaction is the result of meeting the wishes and expectations of the patients. An investigator has developed the Recovery Quality Score-40 (Quality of Recovery Score) and is used to measure the quality of postoperative recovery. This form consists 40 items and is divided into 5 subgroups according to various aspects of the improvement. There are a total of 40 items, 9 related to emotional state, 12 related to physical comfort, 7 related to psychological support, 5 related to physical independence and 7 items related to pain. The questionnaire is scored as a minimum of 40 to a maximum of 200. No special training is required for the implementation of the survey. The fact that the patient can perform the survey on his own and can be done in a short time gives a significant advantage.

The aim of this prospective randomized clinical trial was to compare two different anesthesia applications (sedation & laryngeal mask airway) on anxiety and patient satisfaction in patients with IVF.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) scores of I-II
* Aged 18-55 years old

Exclusion Criteria:

* American Society of Anesthesiology (ASA) scores of III-IV
* Under 18 years of age
* Over 55 years of age,
* Uncontrolled diabetes mellitus, cardiovascular, pulmonary disease, cerebrovascular events,
* Patients with an allergy to anesthetic drugs
* Pregnants
* Patients who refused informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients with In-Vitro Fertilization
Enrollment: 140 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | State-Trait Anxiety Inventory will be performed to the all patients 2 hours before the IVF procedure.
  State-Trait Anxiety Inventory measures state anxiety levels and is an easy-to-implement inventory that the individual can answer on his/her own. The State Anxiety Scale determines how the individual feels himself / herself at a given moment and under certain conditions. It is widely used in preoperative anxiety measurement. State-Trait Anxiety Inventory has 40 items, 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. Responses for the State Anxiety scale assess intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Responses for the Trait Anxiety scale assess frequency of feelings "in general": 1) almost never, 2) sometimes, 3) often, and 4) almost always. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms.
State-Trait Anxiety Inventory | State-Trait Anxiety Inventory will be performed to the all patients 4 hours after the IVF procedure.
  State-Trait Anxiety Inventory measures state anxiety levels and is an easy-to-implement inventory that the individual can answer on his/her own. The State Anxiety Scale determines how the individual feels himself / herself at a given moment and under certain conditions. It is widely used in preoperative anxiety measurement. State-Trait Anxiety Inventory has 40 items, 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. Responses for the State Anxiety scale assess intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Responses for the Trait Anxiety scale assess frequency of feelings "in general": 1) almost never, 2) sometimes, 3) often, and 4) almost always. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms.
Quality of Recovery Score | Quality of Recovery Score will be performed to the all patients 24 hours after the IVF procedure
  Quality of Recovery Score is a global measure of quality of recovery. It incorporates five dimensions of health: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale. Quality of Recovery Scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). This consists 40 items and is divided into 5 subgroups according to various aspects of the improvement. There are a total of 40 items, 9 related to emotional state, 12 related to physical comfort, 7 related to psychological support, 5 related to physical independence and 7 items related to pain. The questionnaire is scored as a minimum of 40 to a maximum of 200.

SECONDARY OUTCOMES:
Heart rate | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Heart rate is measured as beats/minute on the anesthesia monitor
Mean arterial pressure | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Mean arterial pressure is measured as mmHg on the anesthesia monitor
Peripheral oxygen saturation | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Peripheral oxygen saturation is measured as percentage (%) on the anesthesia monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sedat Akbas, Asst. Prof., Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat Akbas, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piroli A, Marci R, Marinangeli F, Paladini A, Di Emidio G, Giovanni Artini P, Caserta D, Tatone C. Comparison of different anaesthetic methodologies for sedation during in vitro fertilization procedures: effects on patient physiology and oocyte competence. Gynecol Endocrinol. 2012 Oct;28(10):796-9. doi: 10.3109/09513590.2012.664193. Epub 2012 Mar 16. PMID 22420562

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03814330/Prot_SAP_000.pdf